CLINICAL TRIAL: NCT05081557
Title: Real World Utilization of Upadacitinib in Adult and Adolescent Patients Living With Moderate to Severe Atopic Dermatitis (AD-VISE)
Brief Title: A Study to Assess Real-World Use, Safety, and Effectiveness of Oral Upadacitinib in Adult and Adolescent (>=12 Years Old) Participants With Atopic Dermatitis
Acronym: AD-VISE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-441
Record Dates: First submitted 2021-10-07; First posted 2021-10-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Atopic Eczema; Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for atopic dermatitis.

SUMMARY:
Atopic dermatitis (AD; also known as atopic eczema) is an inflammatory skin disease. The safety and effectiveness of upadacitinib for AD has been well-documented in previous studies, however, important information is missing on the use patterns and outcomes with upadacitinib in a real-world setting. Therefore, the purpose of this observational study is to help inform real-world usage patterns regarding the safety and effectiveness and duration of response of upadacitinib in adolescent and adult AD participants >=12 years old in the real-world setting.

Upadacitinib is an approved drug being developed for the treatment of AD. Around 975 adolescent and adult participants who are prescribed upadacitinib for the treatment of AD in routine clinical practice will be enrolled worldwide.

Participants will receive oral upadacitinib as prescribed by their physician. Data from these participants will be collected for approximately 2 years.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic and will be asked to provide additional information by questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed diagnosis of atopic dermatitis (AD) or atopic eczema at baseline.
* Symptom onset >=1-year prior to baseline.
* Initiation of upadacitinib treatment for AD is indicated and prescribed per local label.
* The decision to prescribe UPA is made prior to and independently of study participation.
* Medical and medication history available for previous 6 months.
* Participants who can understand the questionnaires, with parental support as required for adolescents.
* Participants who are able to understand and communicate with the investigator and comply with the requirements of the study.
* Participants who are willing and able to participate in the collection of patient-reported data via cloud-based mobile application using a smart device (i.e., tablet).
* Participants who are willing and able to complete the patient-reported questionnaires.

Exclusion Criteria:

- Participants who are currently participating in interventional research (not including non-interventional study, post-marketing observational study, or registry participation).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents (12-17 years of age at baseline) and adults (>=18 years of age at baseline), with a physician-confirmed diagnosis of atopic dermatitis (AD), who are prescribed upadacitinib according to the local label and local practice.
Sampling Method: Non-Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Upadacitinib (UPA) Utilization Patterns | Up to Approximately 24 Months
  UPA utilization patterns will be achieved by (i) providing descriptive statistics of patient demographics and disease characteristics for patients who starting UPA 15 mg at baseline and patients who starting UPA 30 mg at baseline, respectively; (ii) calculating number and proportion of patients with different UPA and concomitant therapy changes throughout the observation period, and the rationale for any changes.
Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) 0/1 | Month 4
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
vIGA-AD 0/1 Among Participants Who Achieved vIGA-AD 0/1 at Month 4 | Month 24
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.

SECONDARY OUTCOMES:
Modification of UPA or Concomitant AD Therapy and Associated Timing, Reasons | Month 24
  This includes UPA dose change, temporary or permanent discontinuation, switching, add or remove TCS.
Percentage of Participants Achieving Eczema Area and Severity Index (EASI) 75 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 90 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 100 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI <=1 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI <=5.9 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI <=7 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving vIGA-AD 0/1 | Up to Approximately 24 Months (Excluding Month 4 - Primary Outcome)
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants Achieving Worst Pruritus Numerical Rating Scale (WP-NRS) 0/1 | Up to Approximately 24 Months
  Worst Pruritus NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving WP-NRS <=3 | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving WP-NRS reduction >=4 | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving Patient Oriented Eczema Measurement (POEM) Score <=2 | Up to Approximately 24 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Percentage of Participants Achieving POEM <=7 | Up to Approximately 24 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID
Percentage of Participants Achieving POEM Reduction >=4 | Up to Approximately 24 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0/1 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving DLQI Score <=5 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving DLQI reduction >=4 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving Atopic Dermatitis Control Tool (ADCT) <7 (control) | Up to Approximately 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess AD control status in adult and adolescent patients (12 years and older). Six AD symptoms and impacts are evaluated over the past week including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions. Each item is scored 0-4. The sum of the 6 item scores form the ADCT total score (range 0-24). A higher score indicates lower AD control. A score of ≥7 indicates that the patient is not in control. The threshold for meaningful within-person change is estimated to be 5 points.
Percentage of Participants Achieving ADCT reduction >=5 | Up to approximately 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess AD control status in adult and adolescent patients (12 years and older). Six AD symptoms and impacts are evaluated over the past week including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions. Each item is scored 0-4. The sum of the 6 item scores form the ADCT total score (range 0-24). A higher score indicates lower AD control. A score of ≥7 indicates that the patient is not in control. The threshold for meaningful within-person change is estimated to be 5 points.
Percentage of Participants who are "Extremely Satisfied" or "Very Satisfied" with their AD Treatment using the Patient Global Impression of Treatment for Atopic Dermatitis (PGIT-AD) | Up to Approximately 24 Months
  PGIT-AD is a single item patient self-administered instrument designed to assess patient satisfaction or dissatisfaction with their current treatment for atopic dermatitis based on the following question: "Overall, how satisfied or dissatisfied are you with your current treatment for atopic dermatitis?". Response options range from 1 (extremely dissatisfied) to 7 (extremely satisfied).
Percentage of Participants Remaining on Upadacitinib Once Daily | Up to Approximately 24 Months
  Percentage of participants remaining on upadacitinib once daily at all applicable time points.
Percentage of Participants Achieving EASI 75 Among Participants Who Achieved EASI 75 at Month 4 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 90 Among Participants Who Achieved EASI 90 at Month 4 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 100 Among Participants Who Achieved EASI 100 at Month 4 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving vIGA-AD 0/1 Among Participants Who Achieved vIGA-AD at Month 4 | Up to Approximately 24 Months (Excluding Month 24 - Primary Outcome)
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants Achieving WP-NRS 0/1 Among Participants Who Achieved WP-NRS 0/1 at Month 4 | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving DLQI Score of 0/1 Among Participants Achieving DLQI Score of 0/1 at Month 4 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving ADCT Reduction <7 Among Participants Who Achieved ADCT Reduction <7 at Month 4 | Up to approximately 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess AD control status in adult and adolescent patients (12 years and older). Six AD symptoms and impacts are evaluated over the past week including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions. Each item is scored 0-4. The sum of the 6 item scores form the ADCT total score (range 0-24). A higher score indicates lower AD control. A score of ≥7 indicates that the patient is not in control. The threshold for meaningful within-person change is estimated to be 5 points.
Absolute Score and Change from Baseline in EASI | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Absolute Score and Change from Baseline in vIGA-AD | Up to Approximately 24 months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Absolute Score and Change from Baseline in Body Surface Area (BSA) | Up to Approximately 24 Months
  The investigator selects the participant's right or left hand as the measuring device. For purposes of clinical estimation, the total surface of the palm plus five digits is assumed to be approximately equivalent to 1%. Measurement of the total area of involvement by the investigator is aided by imagining if scattered plaques were moved so that they were next to each other and then estimating the total area involved. Published score bands: 0% (clear), 0.1-15.9% (mild), 16.0-39.9% (moderate), 40-100% (severe).
Absolute Score and Change from Baseline in WP-NRS | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Absolute Score and Change from Baseline in POEM | Up to Approximately 24 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Absolute Score and Change from Baseline in DLQI | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Absolute Score and Change from Baseline in ADCT | Up to Approximately 24 months
  The ADCT is a validated patient self-administered instrument designed to assess AD control status in adult and adolescent patients (12 years and older). Six AD symptoms and impacts are evaluated over the past week including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions. Each item is scored 0-4. The sum of the 6 item scores form the ADCT total score (range 0-24). A higher score indicates lower AD control. A score of ≥7 indicates that the patient is not in control. The threshold for meaningful within-person change is estimated to be 5 points.
Absolute Score and Change from Baseline in PGIT-AD | Up to Approximately 24 Months
  PGIT-AD is a single item patient self-administered instrument designed to assess patient satisfaction or dissatisfaction with their current treatment for atopic dermatitis based on the following question: "Overall, how satisfied or dissatisfied are you with your current treatment for atopic dermatitis?". Response options range from 1 (extremely dissatisfied) to 7 (extremely satisfied).
Change from Baseline in Flare Frequency and Duration | Up to Approximately 24 Months
  Participants are asked to provide the number of flares in the previous 6 months, and the average duration of flares in the previous 6 months. Participants are asked if currently experiencing an atopic dermatitis flare. Flare is defined as a sudden worsening of AD requiring treatment escalation and/or additional medical advice.
Change from Baseline in the Number of AD-Related Physician Office or Hospital Visits | Up to Approximately 24 Months
  Participants are asked the number of AD-related physician office visits in the previous 6 months and the number of AD-related hospital visits in the previous 6 months.
Absolute Score and Change from Baseline in Work Productivity and Activity Impairment Index for Atopic Dermatitis (WPAI-AD) | Up to Approximately 24 Months
  The Work Productivity and Activity Impairment Index for Atopic Dermatitis (WPAI-AD) is a validated instrument used to measure loss of productivity at work and impairment in daily activities over the past 7 days. The questionnaire includes four items: absenteeism, presenteeism, overall work impairment, and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment. While absenteeism represents the percentage of work time missed due to AD, presenteeism represents the percentage of impairment while at work due to AD. Overall work impairment represents the total percentage of work time missed due to either absenteeism or presenteeism (since those are mutually exclusive). Activity impairment represents the percentage of impairment during daily activities other than work. The 4 items are all evaluated using an 11-point Likert-type scale from 0 (no effect) to 10 (completely prevented), and the scores are multiplied by ten to arrive at a percentage.
Time to Achieve EASI 75 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 90 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 100 | Up to Approximately 24 months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve vIGA-AD 0/1 | Up to Approximately 24 Months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Time to Achieve WP-NRS 0/1 | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Time to Achieve DLQI Score of 0/1 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Time to Achieve POEM <=2 | Up to Approximately 24 Months
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency over the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores (0 to 4) are added to provide a total score range of 0 to 28. The total score reflects disease-related morbidity, and differentiates between "clear/almost clear" (0-2 points), "mild" (3-7 points), "moderate" (8-16 points), "severe" (17-24 points) and "very severe" (25-28 points) AD. A change in POEM score of 3.4 points is considered the MCID.
Time to Achieve ADCT <7 | Up to Approximately 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess AD control status in adult and adolescent patients (12 years and older). Six AD symptoms and impacts are evaluated over the past week including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions. Each item is scored 0-4. The sum of the 6 item scores form the ADCT total score (range 0-24). A higher score indicates lower AD control. A score of ≥7 indicates that the patient is not in control. The threshold for meaningful within-person change is estimated to be 5 points.
Time-Weighted EASI Score | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time-Weighted vIGA-AD Score | Up to Approximately 24 Months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Time-Weighted WP-NRS Score | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Time-Weighted DLQI Score | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving Treatment Target EASI <8 | Up to Approximately 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving Treatment Target DLQI <=5 | Up to Approximately 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Percentage of Participants Achieving Treatment Target WP-NRS <=4 | Up to Approximately 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving Combined Treatment Targets of EASI <8, DLQI <=5, and WP-NRS <=4 | Up to Approximately 24 Months
  EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). DLQI is a 10-item, validated questionnaire to assess the impact of AD disease symptoms and treatment on HRQoL. It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (140):
- Argentina (6):
  - Hospital Universitario Austral /ID# 241607, Pilar, Buenos Aires
  - Buenos Aires Skin /ID# 241606, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - CEDIC Centro de Investigaciones Clinicas /ID# 241605, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia /ID# 241604, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Centro Respiratorio Infantil /ID# 241609, Rosario, Santa Fe Province
  - Hospital Italiano /ID# 241608, CABA
- Australia (6):
  - Kingsway Dermatology & Aesthetics /ID# 242276, Miranda, New South Wales
  - Veracity Clinical Research /ID# 242275, Woolloongabba, Queensland
  - Flinders Medical Centre /ID# 242162, Bedford Park, South Australia
  - Sinclair Dermatology - Melbourne /ID# 242163, East Melbourne, Victoria
  - Burswood Dermatology /ID# 243767, Victoria Park, Western Australia
  - Sydney Skin /ID# 242277, Newtown
- Austria (5):
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 246565, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 247369, Wels, Upper Austria
  - Medizin am Hauptbahnhof /ID# 246567, Vienna, Vienna
  - EZW HAUT Entzuendungszentrum Wien /ID# 246566, Vienna, Vienna
  - Dr. Achim Schneeberger /ID# 247370, Nenzing, Vorarlberg
- Canada (20):
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 240377, Edmonton, Alberta
  - Winnipeg Clinic /ID# 239603, Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc. /ID# 240358, Fredericton, New Brunswick
  - Karma Clinical Trials /ID# 239602, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc. /ID# 239600, St. John's, Newfoundland and Labrador
  - Dr Melinda Gooderham Medicine Profession /ID# 239745, Cobourg, Ontario
  - Dr. Lyne Giroux Medicine Professional Corporation /ID# 240084, Greater Sudbury, Ontario
  - Lima's Excellence in Allergy and Dermatology Research Inc /ID# 239854, Hamilton, Ontario
  - Lynde Institute for Dermatology /ID# 240025, Markham, Ontario
  - Gordon Sussman Medicine Professional Corporation /ID# 243383, North York, Ontario
  - JRB Research /ID# 241862, Ottawa, Ontario
  - Dr. Michael Cecchini Medicine Professional Corporation /ID# 239605, Richmond Hill, Ontario
  - North York Research Inc /ID# 253191, Toronto, Ontario
  - Canadian Dermatology Centre /ID# 240585, Toronto, Ontario
  - Centricity Research - Toronto Dermatology /ID# 241019, Toronto, Ontario
  - Dr Maksym Breslavets Medicine Professional Corporation /ID# 239741, Whitby, Ontario
  - Clinique D /ID# 239601, Laval, Quebec
  - Roula Rassi MD Inc /ID# 252562, Laval, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 239604, Saint-Jérôme, Quebec
  - Clinique de Dermatologie du Haut-Richelieu /ID# 239742, St-Jean Sur Le Richelieu, Quebec
- Czechia (5):
  - Nemocnice Na Bulovce /ID# 246482, Prague, Central Bohemia
  - Nemocnice Ceske Budejovice a.s. /ID# 246479, České Budějovice, Praha 17
  - Fakultni nemocnice Olomouc /ID# 251177, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady /ID# 250792, Prague
  - Duplicate_Fakultni Nemocnice v Motole /ID# 246480, Prague
- Greece (12):
  - Olympion General Clinic /ID# 261694, Pátrai, Achaia
  - Hygeia Hospital /ID# 254188, Amaroussio, Attica
  - 401 GSNA - 401 Army General Hospital /ID# 253222, Athens, Attica
  - 401 GSNA - 401 Army General Hospital /ID# 253228, Athens, Attica
  - University General Hospital Attikon /ID# 253221, Athens, Attica
  - General Hospital Andreas Syggros /ID# 253220, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 253223, Piraeus, Attica
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 253225, Thessaloniki, Evrytania
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 253230, Thessaloniki, Evrytania
  - Papageorgiou General Hospital /ID# 253226, Thessaloniki, Evrytania
  - Naval Hospital of Athens /ID# 253229, Athens
  - University General Hospital of Larissa /ID# 254216, Larissa
- Hungary (5):
  - Semmelweis Egyetem /ID# 239948, Budapest, Budapest
  - Debreceni Egyetem-Klinikai Kozpont /ID# 239949, Debrecen, Hajdú-Bihar
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 239950, Pecs, Nógrád megye
  - Szegedi Tudományegyetem /ID# 239947, Szeged, Szeged
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 239951, Szombathely, Vas County
- Israel (10):
  - Duplicate_Kaplan Medical Center /ID# 244903, Rehovot, Central District
  - Leumit /ID# 260022, Rehovot, Central District
  - HaEmek Medical Center /ID# 247834, Afula, H_efa
  - Rambam Health Care Campus /ID# 244904, Haifa, H_efa
  - Maccabi /ID# 252598, Haifa, H_efa
  - Shaare Zedek Medical Center /ID# 247833, Jerusalem, Jerusalem
  - ZIV Medical Center /ID# 244908, Safed, Northern District
  - The Edith Wolfson Medical Center /ID# 244902, Ashkelon, Southern District
  - Sheba Medical Center /ID# 244905, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 244907, Tel Aviv, Tel Aviv
- Italy (10):
  - A.O.U. Consorziale Policlinico di Bari /ID# 254612, Bari, Bari
  - AOU Policlinico G. Rodolico - San Marco /ID# 255707, Catania, Catania
  - Ospedale San Martino /ID# 255081, Genoa, Genova
  - AOU Gaetano Martino /ID# 255080, Messina, Messina
  - IRCCS Ospedale San Raffaele /ID# 255285, Milan, Milano
  - AOU Citta della Salute e della Scienza di Torino /ID# 254615, Turin, Piedmont
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 255283, Roma, Roma
  - AOU San Giovanni e Ruggi Salerno - Presidio Ospedaliero S.M.I. dell'Olmo /ID# 254689, Cava de' Tirreni, Salerno
  - Azienda ULSS 8 Berica /ID# 255011, Vicenza, Vicenza
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 254613, Novara
- Mexico (12):
  - Centro de Investigacion Biologica y Terapia Avanzada SC (CIMBYTA) /ID# 243820, Guadalajara, Jalisco
  - Centro Dermatologico Del Country S de Rl de Cv /Id# 243818, Guadalajara, Jalisco
  - Grupo Clinico Catei Sociedad Civil /Id# 243809, Guadalajara, Jalisco
  - Consultorio Medico Privado Desiree Larenas Linnemann /Id# 244150, Mexico City, Mexico City
  - Welsh Derm Centro de Especialidades Medicas /Id# 268403, Monterrey, Nuevo León
  - Consultorio Medico Privado Alejandra Macias Weinmann /Id# 244159, Monterrey, Nuevo León
  - Clinica Dermassad /Id# 264048, San Pedro Garza García, Nuevo León
  - Consultorio Medico Privado Cipactli Ariel Navarro Hernandez /Id# 244165, Oaxaca City, Oaxaca
  - Consultorio Medico Privado Yuri Igor Lopez Carrera /Id# 244164, San Andrés Cholula, Puebla
  - Neki Servicios Medicos Profesionales S D Rl de Cv /Id# 243817, Toluca, State of Mexico
  - Consultorio Privado Leslie Lourdes Rodriguez /Id# 243819, Mérida, Yucatán
  - Centro Especializado en Diabetes, Obesidad y Prevencion de Enfermedades Cardiova /ID# 243856, Mexico City
- Poland (6):
  - Maciej Pastuszczak Indywidualna Praktyka Lekarska /ID# 253105, Krakow, Lesser Poland Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny, /ID# 253106, Lublin, Lublin Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 252447, Warsaw, Masovian Voivodeship
  - Prywatna Praktyka Lekarska Witold Owczarek /ID# 252448, Warsaw, Masovian Voivodeship
  - KSW nr1 w Rzeszowie /ID# 251251, Rzeszów, Podkarpackie Voivodeship
  - Dermoklinika Medical Center /ID# 251249, Lodz, Łódź Voivodeship
- Russia (7):
  - Chelyabinsk Regional Clinical Dermatovenerologic Dispensary /ID# 248262, Chelyabinsk, Chelyabinsk Oblast
  - Clinical Dermatovenerology Dispensary /ID# 245225, Krasnodar, Krasnodarskiy Kray
  - Republican hospital named after V.A. Baranov /ID# 245230, Petrozavodsk, Kursk Oblast
  - National Research Center Institute of Immunology of the FMBA of Russia /ID# 245221, Moscow, Moscow
  - Research and Clinical Center for Hematology, Oncology and Immunology, Ryazan Sta /ID# 245220, Ryazan, Ryazan Oblast
  - LLC Scientific Medical Center for General Therapy and Pharmacology /ID# 245229, Stavropol, Stavropol Kray
  - LLC Medical Center ABC of Health /ID# 244816, Kazan', Tatarstan, Respublika
- Spain (20):
  - Hospital Universitario Germans Trias i Pujol /ID# 248512, Badalona, Barcelona
  - Hospital Parc de Salut del Mar /ID# 258675, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 248511, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge /ID# 248513, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Mútua Terrassa /ID# 254292, Terrassa, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 248528, Granada, Granada
  - Hospital Universitario Clinico San Cecilio /ID# 248530, Granada, Granada
  - Hospital Juan Ramon Jimenez /ID# 251960, Huelva, Huelva
  - Hospital Universitario de Jaen /ID# 251959, Jaén, Jaen
  - Hospital San Pedro /ID# 248538, Logroño, La Rioja
  - Hospital Universitario Dr. Negrin /ID# 248533, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Lucus Augusti /ID# 248507, Lugo, Lugo
  - Hospital Universitario Virgen de la Victoria /ID# 248531, Málaga, Malaga
  - Hospital Santa María del Rosell /ID# 251956, Cartagena, Murcia
  - Hospital Universitario de Salamanca /ID# 253356, Salamanca, Salamanca
  - Hospital Universitario Canarias /ID# 251957, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Nuestra Señora de Candelaria /ID# 251961, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocio /ID# 248527, Seville, Sevilla
  - Hospital Clinico Universitario de Valladolid /ID# 253355, Valladolid, Valladolid
  - Hospital Universitario Basurto /ID# 248508, Bilbao, Vizcaya
- Switzerland (7):
  - Kantonsspital Aarau AG /ID# 245517, Aarau, Canton of Aargau
  - Dermatology & Skin Care Clinic /ID# 238348, Buochs, Canton of Nidwalden
  - Kantonsspital St. Gallen /ID# 239244, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich /ID# 240076, Zurich, Canton of Zurich
  - EOC Ospedale Regionale di Bellinzona e Valli /ID# 239246, Bellinzona, Canton Ticino
  - Haut- und Laserzentrum Weinfelden /ID# 239248, Weinfelden, Telangana
  - Basile Darbellay SA /ID# 239245, Orsières, Valais
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 244758, Kaohsiung City, Keelung
  - Chung Shan Medical University Hospital /ID# 244757, Taichung, Keelung
  - National Taiwan University Hospital /ID# 244754, Taipei City, Taipei
  - Chang Gung Memorial Foundation-Taipei Branch /ID# 244760, Taipei
  - Taipei Veterans General Hosp /ID# 244759, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 244756, Taoyuan
- United Arab Emirates (3):
  - New Medical Center Hospital /ID# 245106, Abu Dhabi, Abu Dhabi Emirate
  - Safa Clinic /ID# 248492, Dubai, Dubai
  - Tawam Hospital /ID# 249696, Abu Dhabi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/